CLINICAL TRIAL: NCT00003764
Title: Phase III Randomized Trial of Fludarabine and Cyclophosphamide Versus Fludarabine for Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Fludarabine With or Without Cyclophosphamide in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); SWOG Cancer Research Network (Network)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066890; E2997; CALGB-10103; SWOG-E2997
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known whether combining cyclophosphamide with fludarabine is more effective than fludarabine alone in treating chronic lymphocytic leukemia.

PURPOSE: Randomized phase III trial to study the effectiveness of fludarabine with or without cyclophosphamide in treating patients who have chronic lymphocytic leukemia that has not been treated previously.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of fludarabine with or without cyclophosphamide in terms of complete remission rate and overall survival in patients with previously untreated B cell chronic lymphocytic leukemia (CLL).
* Compare the toxicities of these 2 regimens in this patient population.
* Determine whether the expression of proteins specifically implicated in the regulation of DNA damage induced apoptosis of lymphoid cells (i.e., p53; mdm2; GST; Bcl-2; Mcl-1; Bax; p27; and caspase-3) correlates with response to chemotherapy in these patients.
* Determine whether there is a relationship between clinical response or resistance and differential expression of genes in the CLL cells either at initiation of therapy or following relapse and progression.
* Correlate mutations in immunoglobulin heavy chain variable region genes with clinical response or resistance in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to stage of disease (O-II vs III-IV). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive fludarabine IV over 30 minutes on days 1-5.
* Arm II: Patients receive fludarabine as in arm I plus cyclophosphamide IV over 1 hour on day 1.

Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months until disease progression.

PROJECTED ACCRUAL: A total of 280 patients will be accrued for this study over 2 to 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL) of any stage as defined by the following:

  * Peripheral blood absolute lymphocyte count greater than 5,000/mm^3 within 14 days prior to study
  * Lymphocytes must be small to moderate size with no more than 55% prolymphocytes, atypical lymphocytes, or lymphoblasts morphologically
  * Phenotypically characterized as B-CLL
* Must have one of the following characteristics indicating need for chemotherapy:

  * Progressive marrow failure (hemoglobin less than 10 g/dL and/or platelet count less than 100,000/mm^3)
  * Progressive lymphocytosis with an increase of more than 50% over a 2 month period or anticipated doubling time of less than 6 months
  * Massive (i.e., greater than 6 cm below left costal margin) or progressive splenomegaly
  * Massive nodes or clusters (i.e., greater than 10 cm in longest diameter) or progressive adenopathy
  * At least 10% weight loss within 6 months of study
  * Extreme fatigue
  * Fevers greater than 100.5 degrees F for 2 weeks without evidence of infection
  * Night sweats without evidence of infection
* No autoimmune anemia or autoimmune thrombocytopenia

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2 mg/dL unless secondary to tumor

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 40 mL/min if creatinine is greater than 1.5 mg/dL

Other:

* No other prior or concurrent malignancy within the past 2 years except basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No active infection requiring oral or intravenous antibiotics
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic chemotherapy

Endocrine therapy:

* No prior steroid treatment for CLL

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2000-03-09 (Actual); Primary Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian W. Flinn, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Michael R. Grever, MD, Study Chair — Ohio State University Comprehensive Cancer Center; Mohamad A. Hussein, MD, Study Chair — The Cleveland Clinic
Locations (218):
- United States (215):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Medical Center of Aurora - South Campus, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers - Rose, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Cancer Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Danville Radiation Therapy Center, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- McGill University, Montreal, Quebec, Canada
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Background] Dewald GW, Paietta E, Goloubeva O, et al.: Correlation of interphase fluorescence in situ hybridization (FISH) anomalies with cell morphology and immunophenotyping in chronic lymphocytic leukemia (B-CLL). [Abstract] Blood 100 (11 pt 1): A-2334, 2002.
- [Result] Flinn IW, Neuberg DS, Grever MR, Dewald GW, Bennett JM, Paietta EM, Hussein MA, Appelbaum FR, Larson RA, Moore DF Jr, Tallman MS. Phase III trial of fludarabine plus cyclophosphamide compared with fludarabine for patients with previously untreated chronic lymphocytic leukemia: US Intergroup Trial E2997. J Clin Oncol. 2007 Mar 1;25(7):793-8. doi: 10.1200/JCO.2006.08.0762. Epub 2007 Feb 5. PMID 17283364
- [Result] Grever MR, Lucas DM, Dewald GW, Neuberg DS, Reed JC, Kitada S, Flinn IW, Tallman MS, Appelbaum FR, Larson RA, Paietta E, Jelinek DF, Gribben JG, Byrd JC. Comprehensive assessment of genetic and molecular features predicting outcome in patients with chronic lymphocytic leukemia: results from the US Intergroup Phase III Trial E2997. J Clin Oncol. 2007 Mar 1;25(7):799-804. doi: 10.1200/JCO.2006.08.3089. Epub 2007 Feb 5. PMID 17283363
- [Result] Byrd JC, Gribben JG, Peterson BL, Grever MR, Lozanski G, Lucas DM, Lampson B, Larson RA, Caligiuri MA, Heerema NA. Select high-risk genetic features predict earlier progression following chemoimmunotherapy with fludarabine and rituximab in chronic lymphocytic leukemia: justification for risk-adapted therapy. J Clin Oncol. 2006 Jan 20;24(3):437-43. doi: 10.1200/JCO.2005.03.1021. Epub 2005 Dec 12. PMID 16344317
- [Result] Flinn IW, Kumm E, Grever MR, et al.: Fludarabine and cyclophosphamide produces a higher complete response rate and more durable remissions than fludarabine in patients with previously untreated CLL: Intergroup trial E2997. [Abstract] Blood 104 (11): A-475, 2004.
- [Result] Grever MR, Lucas DM, Dewald GW, et al.: Outcome of treatment with fludarabine versus fludarabine and cyclophosphamide in chronic lymphocytic leukemia (CLL) is adversely impacted by high risk genetic features: results from ECOG 2997. [Abstract] Blood 104 (11 Pt 1): A-3487, 2004.
- [Derived] Lucas DM, Ruppert AS, Lozanski G, Dewald GW, Lozanski A, Claus R, Plass C, Flinn IW, Neuberg DS, Paietta EM, Bennett JM, Jelinek DF, Gribben JG, Hussein MA, Appelbaum FR, Larson RA, Moore DF Jr, Tallman MS, Byrd JC, Grever MR. Cytogenetic prioritization with inclusion of molecular markers predicts outcome in previously untreated patients with chronic lymphocytic leukemia treated with fludarabine or fludarabine plus cyclophosphamide: a long-term follow-up study of the US intergroup phase III trial E2997. Leuk Lymphoma. 2015;56(11):3031-7. doi: 10.3109/10428194.2015.1023800. Epub 2015 Mar 30. PMID 25721902